CLINICAL TRIAL: NCT05248438
Title: Study of Gynecological Follow-up Concerning Women With Multiple Sclerosis
Acronym: GYNESEP
Status: Completed | Type: Observational
Sponsor: University Hospital, Bordeaux (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: CHUBX 2021/49
Record Dates: First submitted 2022-02-11; First posted 2022-02-21 (Actual); Last update posted 2023-06-12 (Actual); Status verified 2023-06

CONDITIONS: Multiple Sclerosis
Keywords: multiple sclerosis; gynecological care; sexuality; contraception
MeSH Terms: conditions — Multiple Sclerosis; Sexuality | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Multiple sclerosis patients: patients affected by multiple sclerosis based on McDonald Criteria 2017
  Interventions: Behavioral: Questionnaire

INTERVENTIONS:
Behavioral: Questionnaire — Questionnaire

SUMMARY:
The investigators want to evaluate gynecological follow-up concerning patients with multiple sclerosis. This study will include reproductive women (from 18 to 40 years old). Patients in the study have an aftercare at the neurology department at Pellegrin Hospital (Bordeaux).

DETAILED DESCRIPTION:
Multiple sclerosis is an inflammatory disease of central nervous system, with a prevalence rate in France of 1 case/1000 subjects (120 000 subjects in France). The average age at diagnosis is 30 years old and it affects especially women, with a sex ratio of 3 women for 1 man.

Many different treatments exist, depending on the severity of the pathology and the evolutivity of the disease. It is very important to understand that some treatments are not compatible with pregnancy. In these circumstances, a regular gynecological follow-up seems to be essential, to discuss contraception and pregnancy. Besides, some treatments have an immunosuppressive activity that is why a gynecological aftercare is necessary, especially in the detection of papillomavirus for cervical cancer.

The neurologist can advise about gynecological issues, but he cannot take care of the gynecological follow-up, that is why it is very interesting to study the quality of the gynecological follow-up. The investigators aim to study gynecological care of patients with multiple sclerosis using a questionnaire made especially for this project. The questionnaire will be filled by patients when they come in the neurology department for a consultation or during their visit at day hospital. At the same time, they will fill a standardized questionnaire about sexuality and quality of life.

This project is a monocentric study realized at Pellegrin Hospital - Bordeaux. Patients with multiple sclerosis belong to a cohort of the neurology center (CRCSEP).

ELIGIBILITY:
Inclusion Criteria:

* Aged between 18 to 40 years old ;
* Diagnosis of multiple sclerosis based on McDonald Criteria 2017 ;
* Patient whose clinical data are referenced in the European Database for Multiple Sclerosis (EDMUS) clinical database (OFSEP database for collecting clinical data from patients followed in the neurology department) ;
* French-speaking, without comprehension disorders ;
* being affiliated to health insurance ;
* Willing to participate and to sign informed consent.

Exclusion Criteria:

* pregnant or breastfeeding women ;
* patient concerned by articles L 1121-5 to L 1121-8 (persons deprived of their liberty by a judicial or administrative decision, minors, persons of legal age who are the object of a legal protection measure or unable to express their consent).

Ages: 18 Years to 40 Years | Sex: Female
Age Groups: Adult
Study Population: Patient Aged between 18 to 40 years old, affected by multiple sclerosis based on McDonald Criteria 2017
Sampling Method: Probability Sample
Enrollment: 192 (Actual)
Dates: Start 2022-05-11 (Actual); Primary Completion 2023-05-09 (Actual); Study Completion 2023-05-09 (Actual)

PRIMARY OUTCOMES:
Gynecological scores of women from 18 to 40 years old with multiple sclerosis with a standardized questionnaire created for the study. | At baseline (Day 0)
  17 questions concerning contraception, number of gynecological follow up, frequency of cervical cancer screening, desire of pregnancy.

SECONDARY OUTCOMES:
Proportion of patients affected by SEP with an Impact on sexuality according to Multiple Sclerosis Intimacy and Sexuality Questionnaire (MSISQ-19). | At baseline (Day 0)
  that varies between 19 and 95 with higher values mean higher levels of Impact on sexuality
Proportion of patients affected by SEP with an impact on life quality according to Fatigue severity Scale (FFS). | At baseline (Day 0)
  that varies between 9 and 63 with higher values mean higher levels of Impact on life quality
Proportion of patients affected by SEP with an impact on life quality according to EHD scores ("échelle d'humeur dépressive" in french) | At baseline (Day 0)
  that varies between 11 and 44 with higher values mean higher levels of Impact on life quality
Proportion of patients affected by SEP with an impact on life quality according to Multiple Sclerosis Quality of life (MusiQol) scores | At baseline (Day 0)
  that varies between 31 and 155 with higher values mean higher levels of Impact on life quality

CONTACTS AND LOCATIONS:
Overall Officials: Valérie BERNARD, MD, Principal Investigator — University Hospital, Bordeaux
Locations (1):
- CHU de Bordeaux - service de neurologie, Bordeaux, France

REFERENCES:
- [Derived] Renaud J, Buissonniere P, Dulau C, Deloire M, Hontarrede F, Montcuquet A, Chansel-Debordeaux L, Hocke C, Ouallet JC, Ruet A, Bernard V. Gynaecological follow-up for women of reproductive age with multiple sclerosis: The GYNESEP study. Mult Scler Relat Disord. 2024 Mar;83:105448. doi: 10.1016/j.msard.2024.105448. Epub 2024 Jan 14. PMID 38277979